CLINICAL TRIAL: NCT05613517
Title: Study of the Correlations Between the Ocular Dominance Depth, the Angle Lambda and the Fixation Disparity in Healthy Individuals
Brief Title: Study of the Angle Lambda and Ocular Dominance
Acronym: EPOLAF
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221023; 2022-A01045-38 (Other: IDRCB Number)
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: No Eye Disorder
Keywords: Angle lambda; Ocular dominance; Fixation disparity; Pupillary axis; Line of sight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy individual: Healthy individual without eye disorder.
  Interventions: Other: Eye examination

INTERVENTIONS:
Other: Eye examination — * orthoptic assessment (visual acuity, refraction, stereopsis test, Cover-test, evaluation of the disparity of fixation and ocular dominance, measurement of the inter-pupillary distance
  * ocular biometry
  * corneal topography
  * monocular photographs in photopic condition

SUMMARY:
Anatomical ophthalmological connections and their dynamics are still debated in the scientific community. However, their considering is essential in many surgeries (strabismus, cataract, refractive...) or in clinical practice.

The correlation between these biometric values would make it possible to refine the knowledge related to these landmarks and thus offer better ophthalmological management by integrating these variables into the clinical examination.

The aim of the study is to analyze the correlation between the angle lambda and the ocular dominance depth in healthy individuals without ophthalmologic disorder.

Then, seconds goals were defined as the study of the relation between the value of the angle lambda and the fixation disparity quantified with the Rousseau test.

Relation between ocular dominance measured with the Guillon's test and the Hole-in-car test will also studied.

DETAILED DESCRIPTION:
The angle lambda corresponds to the angle formed by the pupillary axis (line passing through the center of the pupil and perpendicular to the cornea) and the line of sight (broken line between the fixation point and the fovea and passing through the center of the pupil entrance). The angle kappa corresponds to the angle between the visual axis (line between the point of fixation and the fovea: area of the retina allowing precise vision) and the pupillary axis.

The angle lambda and the angle kappa are very close, which is why the lambda angle is often equated with the kappa angle, both in practice and in the literature.

The literature reports a non-null angle kappa ranged between 1.91° ± 0.14° and 5.73° ± 0.10° in the general population. Also, studies have reported a significantly greater angle on the left eye compared to the right eye. Moreover - because of the interpupillary difference - each eye perceives the same image from a different angle, resulting in a fixation disparity, defined as the angle of the residual deviation of the visual axes when the subject fixes and binocularly merges an image. In some cases, too high a value of the disparity can lead to a fixation disorder requiring orthoptic treatment.

Anatomical ophthalmological connections and their dynamics are still debated in the scientific community. However, their considering is essential in many surgeries (strabismus, cataract, refractive...) or in clinical practice.

The correlation between these biometric values would make it possible to refine the knowledge related to these landmarks and thus offer better ophthalmological management by integrating these variables into the clinical examination.

The aim of the study is to analyze the correlation between the angle lambda and the ocular dominance depth and the fixation disparity in a healthy population without ophthalmologic disorder.

Then, seconds goals were defined as the study of the relation between the value of the angle lambda and the fixation disparity quantified with the Rousseau test.

Relation between ocular dominance measured with the Guillon's test and the Hole-in-car test will also studied.

ELIGIBILITY:
Inclusion Criteria:

- Informed major subject not opposing to their participation in the study

Exclusion Criteria:

* Subject with strabismus or organic ophthalmologic pathology
* Or presenting a visual acuity lower than 10/10th
* Or with a history of eye surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy individuals without visual disorders
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Value of the angle lambda | Day 0
  Semi-automatic digital method of measurement by eye photograph.
Ocular dominance depth | Day 0
  Guillon's and Hole-In-Card tests.

SECONDARY OUTCOMES:
Fixation disparity | Day 0
  Rousseau test.
Ocular dominance measurements quantified by the Hole-in-the-card method | Day 0
  Ocular dominance.
Guillon test | Day 0
  Ocular dominance.
Semi-automatic method of measurement by ocular photography | Day 0
  Compare the values of the lambda angle obtained using the semi-automatic method of measurement by ocular photography and the method using corneal topography.
Method using corneal topography | Day 0
  Compare the values of the lambda angle obtained using the semi-automatic method of measurement by ocular photography and the method using corneal topography.

CONTACTS AND LOCATIONS:
Overall Officials: Maxence Rateaux, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Dominique Bremond-Gignac, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No